CLINICAL TRIAL: NCT02572297
Title: National Network for the Study of Predictors and Prevention of Sudden Unexpected Death in Drug-resistant Partial Epilepsies
Acronym: REPOMSE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2009.582
Record Dates: First submitted 2015-09-04; First posted 2015-10-08 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Drug-resistant Partial Epilepsy
Keywords: epilepsy; SUDEP; SpO2
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- video-EEG: Patients suffering from drug-resistant partial epilepsy for whom a video-EEG monitoring of their seizures was scheduled as part of pre-surgical assessment
  Interventions: Other: video-EEG

INTERVENTIONS:
Other: video-EEG — Registration of seizures during video-EEG

SUMMARY:
Sudden unexpected death in epilepsy (SUDEP) is the main concern of professionals and patient associations involved in epilepsy. These represent a priority for the Ligue Française Contre l'Epilepsie (LFCE). The SUDEP affect primarily young adults, between 18 and 40 years, suffering from epilepsy uncontrolled by medication. In this population of close to 100,000 people in France, the incidence of SUDEP is estimated at 0.5%, or nearly 500 deaths per year. It is clear that the majority of these deaths occur in the immediate consequences of a crisis..

Investigators suppose that a causal link exists between the occurrence of a SUDEP and a per / post-critic decline of SpO2 below 80 % (75 % of cases, 20 % of controls).The constitution of a cohort of 1500 patients clinically well described and a national database will allow other ambitious projects in a speciality where French centres benefit from a unique knowledge, recognized by their foreign colleagues, but underexploited to date. The LFCE (Ligue Française Contre l'Epilepsie) is developing structuring actions to facilitate such exploratory studies for the next two years.

The high death rate which characterizes the drug-resistant partial epilepsies and, in particular, Sudden Unexpected Deaths in Epilepsy (SUDEP) represents the main axis of research for the Ligue Française Contre l'Epilepsie (LFCE) as well as for associations of epileptic patients and the European representatives of the international league against epilepsy ( ILAE). Today, SUDEP occurrences cannot be anticipated. Patients can't be warned against SUDEP.

Although the SUDEP physiopathology remains uncertain, many elements plead for the essential role of a per-and post-critic apnea (central or obstructive). Investigators observe that about 20 % of the patients admitted in a EEG-video monitoring - EEG unit for recording their crisis are going to present experience an per / post-critic severe apnea, severe per / post-critic enough to have induce a SpO2 < 80 % decrease.

However, today, no study has estimated the link relation between the arisen occurrence of such apneas and the later risk of SUDEP.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from drud-resistant partial epilepsy ;
* Patients who are at least 15 years ;
* Patients for whom a video-EEG monitoring of their seizures was scheduled as part of a pre-surgical assessment ;
* Patients having a registration number in the RNIP (Répertoire National d'Identification des Personnes Physiques) or a Social Security number
* Patients who have given their written consent ;
* Patients with a social security

Exclusion Criteria:

* Patients under 15 years
* Patients without drug-resistant partial epilepsy
* Patients without a registration number in the RNIP (Répertoire National d'Identification des Personnes Physiques) or a Social Security number)
* Patient without a consent signed

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from drud-resistant partial epilepsy whom a video-EEG monitoring of their seizures was scheduled as part of a pre-surgical assessment
Sampling Method: Non-Probability Sample
Enrollment: 1072 (Actual)
Dates: Start 2010-05-18 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-08-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with SpO2 < 80% decreases during the EEG-video monitoring | 6 and a half months
  To establish a relation between the occurence of SpO2 < 80% decreases during a EEG-video monitoring and the later risk of SUDEP.

SECONDARY OUTCOMES:
Frequence of other known potential risk factors (composite measure : presence rate of each risk factor in SUDEP measured as percentage) | 6 and a half months
  To test the other potential risk factors of known or still under exploration SUDEPs or still in study (area of the beginning of epilepsy, the abnormalities of sinusal variability). Known potential risk factors are : etiology; epilepsy starting age and duration; crisis frequency in the last 12 months; crisis frequency of secondarly generalized crisis in the last 12 months; presence of nocturnal crisis in the last 12 months; number of concomitant traitments; carbamapezin treatment, Body Mass Indice, sleep apnea syndrome, mood disorder, life qualitity, treatment side effects.
Allelic frequency of genes involved in epileptogenesis (measured as percentage) | 6 and a half months
  Evaluation of the genetic polymorphism of the monoaminergic system or of genes involved in the early epilepsy stage mechanisms of early stages of epilepsy.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe RYVLIN, MD, Principal Investigator — Sercie de neurologie fonctionnelle et d'epileptologie, Hôpital Neurologique Pierre Wertheimer
Locations (1):
- Service de Neurologie Fonctionnelle et d'Epileptologie, Hôpital Pierre Wertheimer, Hospices Civils de Lyon, Bron, France